CLINICAL TRIAL: NCT03856788
Title: Effect of Unilateral Ultrasound-Guided Subcostal Transversus Abdominis Plane Block in Patients Undergoing Laparoscopic Sleeve Gastrectomy
Brief Title: Unilateral TAP Block for Laparoscopic Gastric Sleeve Surgery
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Icahn School of Medicine at Mount Sinai (Other)
Responsible Party: Principal Investigator, Christina Jeng, Associate Professor, Icahn School of Medicine at Mount Sinai
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Other
Other Study IDs: GCO 18-1886
Record Dates: First submitted 2019-02-20; First posted 2019-02-27 (Actual); Results first posted 2022-10-17 (Actual); Last update posted 2022-10-17 (Actual); Status verified 2022-09

CONDITIONS: Laparoscopic Sleeve Gastrectomy; Subcostal Transversus Abdominis Plane Block
Keywords: Randomized control trial; Subcostal transversus abdominis plane block; Laparoscopic sleeve gastrectomy; Regional anesthesia; Opioid consumption; Bariatrics
MeSH Terms: interventions — Sodium Chloride; Bupivacaine

STUDY DESIGN:
Intervention Model Description: The study consists of two study arms. Patients will be getting a subcostal transversus abdominis plane block with either bupivacaine or saline.
Who Masked: Participant, Care Provider, Investigator
Masking Description: Group allocation and instructions on preparing the injectate solution for the subcostal TAP block will be included in a sealed envelope. On the day of the surgery, the group allocation will be revealed to an anesthesiologist not involved with the research study. The anesthesiologist not involved in the study or the care of the patient will prepare the solution to be used for the subcostal TAP block.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (2):
- Saline (Placebo Comparator): Patients will undergo general anesthesia with a post-induction, post-intubation, pre-procedural subcostal TAP block with normal saline on the ipsilateral side as the extraction site.
  Interventions: Drug: Saline
- Bupivacaine (Active Comparator): Patients will undergo general anesthesia with a post-induction, post-intubation, pre-procedural subcostal TAP block with bupivacaine on the ipsilateral side as the extraction site.
  Interventions: Drug: Bupivacaine

INTERVENTIONS:
Drug: Saline — 40 mL sterile normal saline
  Arms: Saline
Drug: Bupivacaine — 40 mL 0.25% bupivacaine
  Arms: Bupivacaine

SUMMARY:
The study team will be assessing if the unilateral subcostal transversus abdominis plane (TAP) block can decrease pain and improve outcomes following laparoscopic sleeve gastrectomy surgeries.

DETAILED DESCRIPTION:
This study will be a double-blinded randomized control trial. Patients will be randomized into one of two groups. Patients in Group 1 will undergo general anesthesia with a post-induction, post-intubation, pre-procedural subcostal TAP block with 40 mL 0.25% bupivacaine on the ipsilateral side as the extraction site. Patients in Group 2 will undergo general anesthesia with a post-induction, post-intubation, pre-procedural subcostal TAP block with 40 mL sterile normal saline on the ipsilateral side as the extraction site. Investigators will be blinded to the randomization of these patients. Following performance of these blocks, patients will receive standard care for the surgery as well as during the postoperative recovery period. Data will be obtained from the EPIC electronic medical record, and from the anesthesia computer record. Patients will be asked postoperatively to assess items such as their nausea and pain scores. Patients will also be contacted by phone within 1-2 days of discharge to obtain analgesic satisfaction scores. This data will be collected on the Redcap server.

ELIGIBILITY:
Inclusion Criteria:

* Adults 18-80 years old
* Candidate for general anesthesia
* Undergoing laparoscopic sleeve gastrectomy
* Patients of participating surgeons

Exclusion Criteria:

* Prior bariatric surgery of any kind
* Previous abdominoplasty
* Allergy or intolerance to one of the study medications
* ASA > 4
* Chronic opioid use (taking opioids for longer than 3 months or daily oral morphine equivalent of >5mg/day for one month)
* History of alcohol/drug abuse
* History of hepatic or renal insufficiency
* Patient refusal

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 43 (Actual)
Dates: Start 2018-12-10 (Actual); Primary Completion 2021-03-25 (Actual); Study Completion 2021-03-25 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Christina Jeng, MD, Principal Investigator — Icahn School of Medicine at Mount Sinai
Locations (1):
- Mount Sinai Brooklyn, New York, New York, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Thorell A, MacCormick AD, Awad S, Reynolds N, Roulin D, Demartines N, Vignaud M, Alvarez A, Singh PM, Lobo DN. Guidelines for Perioperative Care in Bariatric Surgery: Enhanced Recovery After Surgery (ERAS) Society Recommendations. World J Surg. 2016 Sep;40(9):2065-83. doi: 10.1007/s00268-016-3492-3. PMID 26943657
- [Background] Ruiz-Tovar J, Munoz JL, Gonzalez J, Zubiaga L, Garcia A, Jimenez M, Ferrigni C, Duran M. Postoperative pain after laparoscopic sleeve gastrectomy: comparison of three analgesic schemes (isolated intravenous analgesia, epidural analgesia associated with intravenous analgesia and port-sites infiltration with bupivacaine associated with intravenous analgesia). Surg Endosc. 2017 Jan;31(1):231-236. doi: 10.1007/s00464-016-4961-3. Epub 2016 May 13. PMID 27177956
- [Background] Cho JS, Kim HI, Lee KY, Son T, Bai SJ, Choi H, Yoo YC. Comparison of the effects of patient-controlled epidural and intravenous analgesia on postoperative bowel function after laparoscopic gastrectomy: a prospective randomized study. Surg Endosc. 2017 Nov;31(11):4688-4696. doi: 10.1007/s00464-017-5537-6. Epub 2017 Apr 7. PMID 28389801
- [Background] Abdelsalam K, Mohamdin OW. Ultrasound-guided rectus sheath and transversus abdominis plane blocks for perioperative analgesia in upper abdominal surgery: A randomized controlled study. Saudi J Anaesth. 2016 Jan-Mar;10(1):25-8. doi: 10.4103/1658-354X.169470. PMID 26955306
- [Background] Moncada R, Martinaitis L, Landecho M, Rotellar F, Sanchez-Justicia C, Bellver M, de la Higuera M, Silva C, Oses B, Martin E, Perez S, Hernandez-Lizoain JL, Fruhbeck G, Valenti V. Does Preincisional Infiltration with Bupivacaine Reduce Postoperative Pain in Laparoscopic Bariatric Surgery? Obes Surg. 2016 Feb;26(2):282-8. doi: 10.1007/s11695-015-1761-0. PMID 26084250
- [Background] Tsai HC, Yoshida T, Chuang TY, Yang SF, Chang CC, Yao HY, Tai YT, Lin JA, Chen KY. Transversus Abdominis Plane Block: An Updated Review of Anatomy and Techniques. Biomed Res Int. 2017;2017:8284363. doi: 10.1155/2017/8284363. Epub 2017 Oct 31. PMID 29226150
- [Background] McDonnell JG, O'Donnell B, Curley G, Heffernan A, Power C, Laffey JG. The analgesic efficacy of transversus abdominis plane block after abdominal surgery: a prospective randomized controlled trial. Anesth Analg. 2007 Jan;104(1):193-7. doi: 10.1213/01.ane.0000250223.49963.0f. PMID 17179269
- [Background] Shibata Y, Sato Y, Fujiwara Y, Komatsu T. Transversus abdominis plane block. Anesth Analg. 2007 Sep;105(3):883; author reply 883. doi: 10.1213/01.ane.0000268541.83265.7d. No abstract available. PMID 17717265
- [Background] Lee TH, Barrington MJ, Tran TM, Wong D, Hebbard PD. Comparison of extent of sensory block following posterior and subcostal approaches to ultrasound-guided transversus abdominis plane block. Anaesth Intensive Care. 2010 May;38(3):452-60. doi: 10.1177/0310057X1003800307. PMID 20514952
- [Background] Ari DE, Ar AY, Karip CS, Koksal C, Aydin MT, Gazi M, Akgun F. Ultrasound-guided subcostal-posterior transversus abdominis plane block for pain control following laparoscopic sleeve gastrectomy. Saudi Med J. 2017 Dec;38(12):1224-1229. doi: 10.15537/smj.2017.12.21133. PMID 29209672
- See also: Subcostal TAP Block — https://www.nysora.com/ultrasound-guided-transversus-abdominis-plane-quadratus-lumborum-blocks

RESULTS

PARTICIPANT FLOW:
Groups:
- Saline: Patients underwent general anesthesia with a post-induction, post-intubation, pre-procedural subcostal Transversus Abdominis Plane (TAP) block with normal saline on the ipsilateral side as the extraction site.
  Saline: 40 mL sterile normal saline
- Bupivacaine: Patients underwent general anesthesia with a post-induction, post-intubation, pre-procedural subcostal TAP block with bupivacaine on the ipsilateral side as the extraction site.
  Bupivacaine: 40 mL 0.25% bupivacaine
Period: Overall Study
Arm/Group | Saline | Bupivacaine
Started | 23 | 20
Completed | 21 | 19
Not Completed | 2 | 1

BASELINE CHARACTERISTICS:
Groups:
- Saline: Patients underwent general anesthesia with a post-induction, post-intubation, pre-procedural subcostal TAP block with normal saline on the ipsilateral side as the extraction site.
  Saline: 40 mL sterile normal saline
- Total: Total of all reporting groups
Arm/Group | Saline | Bupivacaine | Total
Number analyzed (Participants) | 21 | 19 | 40
Age, Continuous [Median (Inter-Quartile Range); unit: years] | 40 [32 to 43] | 36 [29 to 45.5] | 36.5 [31 to 43]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 9 | 16 | 25
  Male | 12 | 3 | 15
Race and Ethnicity Not Collected [Count of Participants; unit: Participants] — Population: Race and Ethnicity were not collected from any participant.

OUTCOME MEASURES:

1. Primary Outcome: Amount of 24 Hour Opioid Consumption
Description: Amount of intravenous (IV) opioid consumption within 24-hour period
Time Frame: 24 Hours postoperative
Measure: Median (Inter-Quartile Range); unit: morphine milligram equivalents
Arm/Group | Saline | Bupivacaine
Number analyzed (Participants) | 21 | 19
morphine milligram equivalents | 44.7 [33.4 to 59.8] | 38.7 [24 to 49]

2. Secondary Outcome: Amount of Intraoperative IV Opioid Consumption
Description: Amount of intravenous opioid consumption during the surgery
Time Frame: average 2-3 Hours
Measure: Median (Inter-Quartile Range); unit: morphine milligram equivalents
Arm/Group | Saline | Bupivacaine
Number analyzed (Participants) | 21 | 19
morphine milligram equivalents | 35 [32.5 to 40] | 32.5 [25 to 447.5]

3. Secondary Outcome: Number of Participants Asked Area of Pain on the Body After Surgery
Description: Patients asked for the areas of pain (right upper quadrant (RUQ), left upper quadrant, (LUQ) right lower quadrant (RLQ), or left lower quadrant (LLQ), diffuse and epigastric) after surgery.
Time Frame: 24 Hours postoperative
Measure: Count of Participants; unit: Participants
Arm/Group | Saline | Bupivacaine
Number analyzed (Participants) | 21 | 19
Participants
  none | 3 | 7
  diffuse | 7 | 1
  RUQ | 3 | 3
  LUQ | 1 | 2
  RLQ | 0 | 0
  LLQ | 0 | 0
  epigastric | 7 | 6

4. Secondary Outcome: Number of Participants Who Answered Yes to Having Presence of Nausea After Surgery
Description: Number of participants who answered yes to having presence of nausea after surgery
Time Frame: 24 Hours postoperative
Measure: Count of Participants; unit: Participants
Arm/Group | Saline | Bupivacaine
Number analyzed (Participants) | 21 | 19
Participants | 16 | 14

ADVERSE EVENTS:
Time Frame: 1 year postoperative
Description: Participants followed at one year postoperative for mortality.
Arm/Group | Saline | Bupivacaine
All-Cause Mortality (participants affected / at risk) | 0/23 | 0/20
Serious Adverse Events (participants affected / at risk) | 0/23 | 0/20
Other Adverse Events (participants affected / at risk) | 0/23 | 0/20

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (3):
  • Study Protocol (2019-09-09): https://cdn.clinicaltrials.gov/large-docs/88/NCT03856788/Prot_000.pdf
  • Statistical Analysis Plan (2022-08-24): https://cdn.clinicaltrials.gov/large-docs/88/NCT03856788/SAP_001.pdf
  • Informed Consent Form (2019-10-09): https://cdn.clinicaltrials.gov/large-docs/88/NCT03856788/ICF_002.pdf